CLINICAL TRIAL: NCT06567925
Title: Sleep Extension to Improve Sleep Efficiency and Quality of Life in Heart Failure With Preserved Ejection Fraction: the SLEEP-HF Pilot Study
Brief Title: Sleep Extension to Improve Sleep Efficiency and QoL in HF With Preserved Ejection Fraction: the SLEEP-HF Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Sleep Research Society Foundation (SRSF) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20028346
Record Dates: First submitted 2024-08-01; First posted 2024-08-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Sleep Efficiency; Sleep Extension; Heart Failure with Preserved Ejection Fraction; Quality of Life

STUDY DESIGN:
Intervention Model Description: Single-arm open-label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gradual sleep extension strategy (Experimental): Demonstrate the feasibility of a gradual sleep extension strategy combined with sleep hygiene training aimed at increasing sleep efficiency in patients with heart failure with preserved ejection fraction on guideline-directed medical therapy
  Interventions: Behavioral: Customized Sleep Coaching; Behavioral: Sleep Hygiene Training

INTERVENTIONS:
Behavioral: Customized Sleep Coaching — Demonstrate the feasibility of a gradual sleep extension strategy using customized sleep coaching.
Behavioral: Sleep Hygiene Training — Sleep hygiene training aimed at increasing sleep efficiency in patients with heart failure with preserved ejection fraction on guideline-directed medical therapy

SUMMARY:
Nearly one-third of US adults have poor sleep quality. Sleep quality refers to sleep efficiency, sleep latency, sleep duration, wake after sleep onset, and movement during the night. Specifically, sleep efficiency (SE) measures how well an individual utilizes their time in bed for restorative sleep and it highly depends on actual sleep duration. Reduced SE is associated with a greater risk for heart failure (HF), which affects ~6.7 million adults in the US alone. HF with preserved ejection fraction (HFpEF) accounts for about half of all HF diagnoses and is associated with poor prognosis (30-50% 5-year mortality from diagnosis) and severely reduced quality of life (QoL). Long-term goal for the investigators is to identify sleep modulation as a potential therapeutic target to improve QoL in HFpEF, with poor SE being present in ~60% of patients with HFpEF. The study is aimed to see if the sleep modulation is feasible and modulating sleep can improve the QoL and functional capacity along with the reduction of inflammation among subjects with HFpEF.

DETAILED DESCRIPTION:
The investigators plan a 2-week single-arm open-label feasibility study in 17 subjects with HFpEF with a 1-week run-in phase (3 weeks total duration) with a sleep extension intervention combined with sleep hygiene training to improve SE in patients with symptomatic HFpEF. The investigator's primary endpoint is to increase sleep duration and efficiency with this intervention.

ELIGIBILITY:
Inclusion Criteria:

* confirmed clinical diagnosis of stable HF (NYHA class II-III)
* left ventricular ejection fraction>50% documented in the prior 12 months
* aged ≥18 years
* habitual reported sleep duration ≤7 hours
* sleep efficiency <85% measured during the 1-week run-in phase

Exclusion Criteria:

* concomitant conditions that can limit physical activity
* severe debilitating diseases (ischemic heart disease. angina, arterial fibrillation, moderate to severe valvular disease)
* taking sleep medicine or melatonin irregularly
* pregnancy
* stage V kidney disease (with dialysis)
* shift worker
* insomnia
* hospitalization within the last 2 months
* patients with sleep and circadian disorders
* fluid overload
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate the feasibility of a gradual sleep extension strategy combined with sleep hygiene training using a wearable device | Between baseline and 2 weeks of the intervention
  To assess the sleep modulation, We will assess sleep quality using the two wearable devices. A research-based accelerometer (GT9X Link, ActiGraph, FL) will be used on the wrist using a 24-hour per day for 7 days wear protocol except shower and swimming for the 1-week run-in phase. The same wear protocol will be implemented for the 2 weeks of intervention. Sleep duration and rest in bed will be automatically detected by the Actigraph and translated by Actilife software with an epoch of 30 seconds.
Demonstrate the feasibility of a gradual sleep extension strategy combined with sleep hygiene training using a sleep journal | Between baseline and 2 weeks of the intervention
  A sleep diary will be used to reinforce the assessment conducted by accelerometer. A sleep diary is a record of your sleep behaviors, quality and schedule. It can help you to gauge your total sleep time, mark your breaks in sleep and when they occur and track changes in your quality of sleep.
Demonstrate the feasibility of a gradual sleep extension strategy combined with sleep hygiene training using the Pittsburgh Sleep Quality questionnaire. | Baseline (week 1) and at the end of the follow-up period (week 3)
  Pittsburgh Sleep Quality questionnaire: Pittsburgh Sleep Symptom Questionnaire - Insomnia (PSSQ_I) has 13 self-rated questions. Only questions 1,2 or 5 are used to determine the presence, frequency AND duration of sleep symptom criteria. Questions 6-13 are used to identify significant daytime consequences of the sleep complaint. Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep
Demonstrate the feasibility of a gradual sleep extension strategy combined with sleep hygiene training using the Epworth Sleepiness Scale at baseline and at the end of the follow-up for subjectively assess sleep quality. | Baseline (week 1) and at the end of the follow-up period (week 3)
  Epworth Sleepiness Scale: The Epworth sleepiness scale results range from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness. A result under 10 may not be cause for concern or it could identify you have trouble sleeping (insomnia). A result from 11 to 24 indicates excessive (abnormal) daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Carbone, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States